CLINICAL TRIAL: NCT01308424
Title: A Randomized, Double-blind, Parallel, Placebo-controlled Study for the Assessment of the Safety and Efficacy of BTL-TML-HSV for the Treatment of Recurrent Symptomatic Oral Herpes Virus Infection
Brief Title: Safety and Efficacy Study of a New Treatment for Recurrent Symptoms of Oral Herpes Virus Infection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beech Tree Labs, Inc. (Industry)
Collaborators: Norwich Clinical Research Associates Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010-03-0112
Record Dates: First submitted 2011-03-02; First posted 2011-03-04 (Estimated); Results first posted 2013-08-13 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Oral Herpes Simplex
Keywords: Herpes Labialis; Herpes Simplex; Herpes
MeSH Terms: conditions — Stomatitis, Herpetic; Herpes Labialis; Herpes Simplex

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BTL TML HSV (Experimental)
  Interventions: Drug: BTL TML HSV
- Matching Placebo (Placebo Comparator)
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: BTL TML HSV — Sublingual micro-dosing for 7 days
  Arms: BTL TML HSV
Drug: Matching placebo — sublingual dosing for 7 days
  Arms: Matching Placebo

SUMMARY:
The purpose of this study is to determine if a new treatment is effective for the treatment of recurrent symptomatic oral herpes virus infections.

ELIGIBILITY:
Inclusion Criteria:

* Clinical history of recurrent cold sores averaging 2 or more episodes per year
* Experiences prodromal symptoms (tingling, burning, itching) of cold sores
* Herpes Simplex Virus seropositive (by blood test)

Exclusion Criteria:

* Immuno-suppressed or taking immunosuppressant medication
* Use of antiviral therapy directly prior and during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2011-01; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Kentucky College of Dentistry/Center for Oral Health Research, Lexington, Kentucky
  - School of Dental Medicine, University at Buffalo, Buffalo, New York
  - Family Dentistry, Norwich, New York
  - University of Pittsburgh School of Dental Medicine, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Mamber SW, Hatch T, Miller CS, Murray JV, Strout C, McMichael J. Low-dose Oral Thimerosal for the Treatment of Oral Herpes: Clinical Trial Results and Improved Outcome After Post-hoc Analysis. J Evid Based Integr Med. 2022 Jan-Dec;27:2515690X221078004. doi: 10.1177/2515690X221078004. PMID 35142535

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from four dental clinics in the USA during the study period of 1/26/11 - 9/14/2012
Pre-assignment Details: Participants entered a baseline run in period to assess eligibility before randomization and dental procedure.
Groups:
- Baseline Run In: Baseline period to assess eligibility before randomization
- Matching Placebo: Matching placebo : sublingual dosing for 7 days
- BTL TML HSV: BTL TML HSV : Sublingual micro-dosing for 7 days
Period: Baseline Eligibility
Arm/Group | Baseline Run In | Matching Placebo | BTL TML HSV
Started | 242 | 0 | 0
Completed | 171 (Completed baseline run in and were eligible for randomization) | 0 | 0
Not Completed | 71 | 0 | 0
Not completed — Screen Failures | 71 | 0 | 0
Period: Randomization
Arm/Group | Baseline Run In | Matching Placebo | BTL TML HSV
Started | 0 | 87 | 84
Completed | 0 | 84 | 82
Not Completed | 0 | 3 | 2
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Subjects randomized into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Matching Placebo | BTL TML HSV | Total
Number analyzed (Participants) | 87 | 84 | 171
Age Continuous [Mean (Full Range); unit: years] | 41.6 [19.2 to 70.7] | 45.2 [20.0 to 76.9] | 43.3 [19.2 to 76.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 61 | 116
  Male | 32 | 23 | 55
Region of Enrollment [Number; unit: participants]
  United States | 87 | 84 | 171

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Who Experience a New Cold Sore Outbreak That Proceeds to the Lesion Stage. Of Those Subjects That Take Study Medication (Experience a New Emerging Cold Sore) Those That Proceed to Lesion Stage (Cold Sore Stage - 3 Vesicle or Above).
Description: Subjects start a daily diary based on start of symptoms of a new emerging cold sore and start taking study medication. Subjects note the start time of study medication along with cold sore stage(s)for at least 7 days and up to 14 days. Subjects take study medication for 7 days. Cold Sore stages are 0=Dormant, 1=Prodrome, 2=Inflammation, 3=Vesicle, 4=Ulcer, 5=Crust, 6=Healed. If subjects do not experience a new cold sore outbreak within 7 days, they do not take study medication and are completed with the study.
Time Frame: 7-14 days (depending on time of lesion outbreak - subjects had 7 days to experience a new emerging cold sore)
Population: As randomized subjects waited until reoccurrence of cold sore lesions, 23/87 participants in the placebo treatment group and 9/84 in the BTL-TML-HSV group took study medication and were eligible for the primary outcome.
Measure: Number; unit: percentage of Participants
Arm/Group | Matching Placebo | BTL TML HSV
Number analyzed (Participants) | 23 | 9
percentage of Participants | 77.8 | 45.5

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the time of signing informed consent till the subjects completed the study (up to 28 days)
Description: Adverse Events were assessed at each study visit, and from subject diary.
Arm/Group | Baseline Run In | Matching Placebo | BTL TML HSV
Serious Adverse Events (participants affected / at risk) | 0/71 | 2/87 | 0/84
Other Adverse Events (participants affected / at risk) | 0/71 | 32/87 | 29/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baseline Run In (N=71) | Matching Placebo (N=87) | BTL TML HSV (N=84)
Post Colonoscopy bowel perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Subject developed complications during a routine colonoscopy procedure
Low Blood Volume (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baseline Run In (N=71) | Matching Placebo (N=87) | BTL TML HSV (N=84)
Headache (Nervous system disorders) | 0 (0) | 7 (10) | 9 (11)
Oral lesion (Gastrointestinal disorders) | 0 (0) | 6 (7) | 1 (1)
High protein urine (Investigations) | 0 (0) | 7 (7) | 4 (4) — Labs could have been taken at baseline prior to randomization.
High Red Blood Cells urine (Investigations) | 0 (0) | 5 (5) | 6 (6) — Labs could have been taken at baseline prior to randomization.
Urine ketone body (Investigations) | 0 (0) | 5 (5) | 4 (4) — Labs could have been taken at baseline prior to randomization.
Urine White Blood Cells (Investigations) | 0 (0) | 2 (2) | 5 (5) — Labs could have been taken at baseline prior to randomization.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days